CLINICAL TRIAL: NCT06594718
Title: Endoscopic Treatment of Zenker's Diverticulum: a Prospective Observational Study Comparing Tunnelization (Z-POEM) Versus Non-Tunnelization Techniques
Brief Title: Endoscopic Treatment of Zenker's Diverticulum (ZENKTUN)
Status: Not yet recruiting | Type: Observational
Sponsor: Société Française d'Endoscopie Digestive (Other)
Responsible Party: Principal Investigator, Bertrand Brieau, Medical doctor, Principal Investigator, Société Française d'Endoscopie Digestive
Other Study IDs: SFED 157
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Zenker Diverticulum
Keywords: Zenker's diverticulum; Z-POEM; Diverticuloscope; Knife Septotomy; Clutch Cutter
MeSH Terms: conditions — Zenker Diverticulum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Endoscopic treatment with (Z-POEM): Patients undergoing a peroral endoscopic myotomy using a tunneling method to access the target zone.
  Interventions: Procedure: Endoscopic diverticulotomy with Z-POEM
- Endoscopic treatment using a non-tunnelization technique: Patients undergoing a peroral endoscopic myotomy using a no-tunneling method (Diverticuloscope, Knife Septotomy, and Clutch Cutter) to access the target zone.
  Interventions: Procedure: Endoscopic diverticulotomy using a non-tunnelization technique

INTERVENTIONS:
Procedure: Endoscopic diverticulotomy with Z-POEM — Endoscopic diverticulotomy with Z-POEM
  Groups: Endoscopic treatment with (Z-POEM)
Procedure: Endoscopic diverticulotomy using a non-tunnelization technique — Endoscopic diverticulotomy with diverticuloscope, Knife Septotomy, or Clutch Cutter
  Groups: Endoscopic treatment using a non-tunnelization technique

SUMMARY:
Prospective comparative observational study in numerous reference centers in France, comparing Tunnelization (Z-POEM) versus Non-Tunnelization Techniques according to the usual practices. This is a prospective, comparative, observational, multicenter study with the primary objective of comparing the symptomatic recurrence rate one year after endoscopic tunnelization therapy (Z-POEM) versus non-tunnelization techniques in patients with symptomatic Zenker's diverticulum.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic Zenker's diverticulum (Augsburg score ≥5 )
* Diagnostic evaluation including esophagogastroduodenoscopy (EGD) and a barium swallow (TOGD) with measurement of the diverticulum's height.
* Patient aged 18 years or older
* Patient with ASA 1, ASA 2, ASA 3 status
* No participation in another concurrent clinical study

Exclusion Criteria:

* Patient under 18 years old
* Patient with ASA 4 or ASA 5 status
* Pregnant woman
* Patient with coagulation disorders preventing the performance a polypectomy: PT < 50%, Platelets < 50,000/mm³, ongoing effective anticoagulation, or current clopidogrel use.
* Patient who has already undergone initial endoscopic or surgical treatment for Zenker's diverticulum

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient referred for endoscopic treatment of symptomatic Zenker's diverticulum
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2024-10-31 (Estimated); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Symptomatic recurrence rate after endoscopic tunnelization therapy (Z-POEM) compared to non-tunnelization techniques in patients with symptomatic Zenker's diverticulum. | 12 months
  Symptomatic recurrence is defined by:
  Clinical resolution after endoscopic treatment, as assessed clinically at 3 months, with an Augsburg score <5.
  Reappearance of clinical symptoms, following clinical resolution after endoscopic treatment, with an Augsburg score ≥5.

SECONDARY OUTCOMES:
Clinical success rate after endoscopic treatment. | 3 months
  Clinical success is assessed using the Augsburg scale, with a score <5.
Variation in Augsburg score at different time points | 3 months, 6 months, 12 months, and 24 months
  comparing the Augsburg scores at each time point with baseline data for each patient.
Complication rate associated with the endoscopic procedure | 15 days
  Number of patients with at least one of the following complications: Pneumoperitoneum insufflation, Fever during hospitalization (T > 38.5°C), Post-procedure hemorrhage, Post-procedure antibiotic therapy, Post-procedure scan, Intensive care unit/rehabilitation hospitalization, or Surgery for complications
Radiographic resolution rate of the diverticulum | 3 months
  Radiographic resolution rate of the diverticulum, assessed by a TOGD (barium swallow) at 3 months: Radiographic resolution is defined by a reduction in the diverticulum's volume between the preoperative TOGD and the TOGD at 3 months. The volume is estimated from the millimeter measurements of the diverticulum in its craniocaudal, anteroposterior, and laterolateral dimensions. The definitions are as follows:
  Complete resolution: Complete disappearance of the diverticulum. Partial resolution: Reduction in diverticular volume of at least 50%. Minor resolution: Reduction in diverticular volume between 20% and 50%. No resolution: Reduction in diverticular volume < 20%.
Symptomatic Recurrence Rate Post-Treatment: | at 3, 6, 12, and 24 Months
  Number of patients with symptomatic recurrence, defined as the reappearance of clinical symptoms at 3, 6, 12, and 24 months after endoscopic treatment, with an Augsburg score of ≥5.

IPD SHARING:
Plan to Share IPD: No